CLINICAL TRIAL: NCT05223283
Title: Limb Salvage Related to Venous Injury: Case Series
Brief Title: Limb Salvage Post Venous Injury:Case Series
Status: Completed | Type: Observational
Sponsor: Jabir Ibn Hayyan Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Limb salvage
Record Dates: First submitted 2021-10-18; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2021-10

CONDITIONS: Limb Salvage
Keywords: limb salvage; venous injury; edema; amputation; fasciotomy.
MeSH Terms: conditions — Edema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
The venous injury diagnosis depends on history of trauma with symptoms and signs suggestive of venous injuries and color flow duplex study is of increasing value as a screen for detection of an occult venous injuries. It is associated with arterial, peripheral nerve injuries and bone fractures. Within this study of one-year duration, a seventy-five patients with acute venous injuries were included. The injured vein was either repaired or ligated according to hemodynamic state of patient and site and type of injury.

DETAILED DESCRIPTION:
This is a retrospective cross section study of one-year duration from January 2017 and January 2019 at Najaf Teaching medical city/Iraq . The study included a Seventy-five patients with acute venous injuries. The Venous surgical interference for late complicated vascular injuries and iatrogenic venous injuries were excluded and the information was obtained from the hospital records and direct evaluation of patients.

ELIGIBILITY:
Inclusion Criteria:

All in surgical emergency departments

Exclusion Criteria:

nil

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All limb injured patient
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Limb salvage or amputation | two years
  Venous limb injury

IPD SHARING:
Plan to Share IPD: Undecided